CLINICAL TRIAL: NCT05338775
Title: A Phase 1b Study of Bispecific T Cell Redirection Antibodies in Combination With Checkpoint Inhibition for the Treatment of Participants With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of Talquetamab and Teclistamab Each in Combination With a Programmed Cell Death Receptor-1 (PD-1) Inhibitor for the Treatment of Participants With Relapsed or Refractory Multiple Myeloma
Acronym: TRIMM-3
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR109168; 64407564MMY1005 (Other: Janssen Research & Development, LLC); 2021-005073-22 (EudraCT Number); 2022-502681-24-00 (Registry Identifier: EUCT number)
Expanded Access: NCT05503550 (No longer available)
Record Dates: First submitted 2022-03-31; First posted 2022-04-21 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Relapsed/ Refractory Multiple Myeloma
MeSH Terms: interventions — talquetamab; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): Participants will receive either talquetamab (treatment regimen A) or teclistamab (treatment regimen B) with a PD-1 inhibitor biweekly.
  Interventions: Drug: Talquetamab; Drug: Teclistamab; Drug: PD-1 Inhibitor
- Part 2: Dose Expansion (Experimental): Participants will receive either treatment regimen A or treatment regimen B with a PD-1 inhibitor at the dose levels identified in Part 1.
  Interventions: Drug: Talquetamab; Drug: Teclistamab; Drug: PD-1 Inhibitor

INTERVENTIONS:
Drug: Talquetamab — Talquetamab will be administered as a subcutaneous (SC) injection.
Drug: Teclistamab — Teclistamab will be administered as a SC injection.
Drug: PD-1 Inhibitor — The PD-1 inhibitor will be administered as an intravenous injection.

SUMMARY:
The purpose of the study is to identify the safe dose(s) of a PD-1 inhibitor in combination with talquetamab or teclistamab, and to characterize the safety and tolerability of talquetamab or teclistamab when administered in combination with a PD-1 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Have documented initial diagnosis of multiple myeloma according to International Myeloma Working Group (IMWG) diagnostic criteria
* Participants with relapsed or refractory disease that are not a candidate for available therapy with established clinical benefit
* Have measurable disease at screening as defined by at least 1 of the following: a) Serum M-protein level greater than or equal to (>=) 0.5 grams per deciliter (g/dL); b) Urine M-protein level >= 200 milligrams (mg) per 24 hours; c) Light chain multiple myeloma: Serum immunoglobulin (Ig) free light chain (FLC) >= 10 milligrams/deciliter (mg/dL) and abnormal serum Ig kappa lambda FLC ratio
* Have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1

Exclusion Criteria:

* Prior antitumor therapy within 21 days prior to the first dose of study treatment (proteasome inhibitor [PI] therapy or radiotherapy within 14 days, immunomodulatory drug (IMiD) agent therapy within 7 days, gene -modified adoptive cell therapy or autologous stem cell transplant within 3 months)
* Prior therapy with PD-1 inhibitors, allogeneic stem cell transplant or solid organ transplant
* Active plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, M-protein, and skin changes), or primary light chain amyloidosis
* Active Central Nervous System (CNS) involvement or exhibition of clinical signs of meningeal involvement of multiple myeloma. If either is suspected, brain magnetic resonance imaging (MRI) and lumbar cytology are required
* Live, attenuated vaccine within 4 weeks before the first dose of study treatment
* Non-hematologic toxicity from prior anticancer therapy that has not resolved to baseline levels or to Grade less than or equal to (<=) 1 (except alopecia [any grade] or peripheral neuropathy to Grade <= 2)
* Received a cumulative dose of corticosteroids equivalent to >= 140 milligrams (mg) of prednisone within the 14-day period before the start of study treatment administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2027-05-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 2 years 5 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with Adverse Events (AEs) by Severity | Up to 2 years 5 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening, and Grade 5= Death related to adverse event.
Number of Participants with Abnormalities in Clinical Laboratory Assessments | Up to 2 years 5 months
  Number of participants with abnormalities in clinical laboratory assessments (serum chemistry and hematology) will be reported.
Number of Participants with Dose-Limiting Toxicity (DLTs) | Up to 2 years 5 months
  The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 2 years 5 months
  ORR is defined as the percentage of participants who achieve partial response (PR) or better according to the International Myeloma Working Group (IMWG) 2016 criteria.
Very Good Partial Response (VGPR) or Better Response Rate | Up to 2 years 5 months
  VGPR or better response rate is defined as the percentage of participants who achieve a VGPR or better response (stringent complete response [sCR]+ complete response [CR]+VGPR) according to the IMWG 2016 criteria.
Complete Response (CR) or Better Response Rate | Up to 2 years 5 months
  CR or better response rate is defined as the percentage of participants who achieve a CR or better response (sCR+CR) according to the IMWG 2016 criteria.
Stringent Complete Response (sCR) Rate | Up to 2 years 5 months
  sCR rate is defined as the percentage of participants who achieve an sCR according to the IMWG 2016 criteria.
Duration of Response | Up to 2 years 5 months
  Duration of response is defined as time from date of initial documentation of a response (PR or better) to date of first documented evidence of progressive disease (PD), per IMWG 2016 criteria or death due to any cause, whichever occurs first.
Time to Response | Up to 2 years 5 months
  Time to response is defined as the time between date of first dose of study treatment and the first efficacy evaluation at which the participant has met all criteria for PR or better.
Serum Concentrations of Talquetamab | Up to 2 years 5 months
  Serum samples will be analyzed to determine concentrations of Talquetamab using validated, specific, and sensitive immunoassay methods.
Serum Concentrations of Teclistamab | Up to 2 years 5 months
  Serum samples will be analyzed to determine concentrations of Teclistamab using validated, specific, and sensitive immunoassay methods.
Serum Concentrations of PD-1 Inhibitor | Up to 2 years 5 months
  Serum samples will be analyzed to determine concentrations of PD-1 inhibitor using validated, specific, and sensitive immunoassay methods.
Number of Participants with Anti-Talquetamab Antibodies | Up to 2 years 5 months
  Number of participants with anti-talquetamab antibodies will be reported.
Number of Participants with Anti-Teclistamab Antibodies | Up to 2 years 5 months
  Number of participants with anti-teclistamab antibodies will be reported.
Number of Participants with Anti-PD-1 Inhibitor Antibodies | Up to 2 years 5 months
  Number of participants with anti-PD-1 inhibitor antibodies will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research and Development, LLC Clinical Trial, Study Director — Janssen Research and Development LLC
Locations (19):
- United States (7):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - The Blavatnik Family Chelsea Medical Center at Mount Sinai, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
- France (4):
  - CHU de Montpellier Hopital Saint Eloi, Montpellier
  - CHU de Nantes hotel Dieu, Nantes
  - CHU Poitiers - Hopital la Miletrie, Poitiers
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
- Germany (4):
  - Universitatsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitatsklinikum Wurzburg, Würzburg
- Spain (4):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp Clinico Univ de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency